CLINICAL TRIAL: NCT03746639
Title: Effects of Therapeutic Ultrasound Applied to The Lumbar Region on Renal Function: A Randomised Controlled Prospective Trial
Brief Title: Therapeutic Ultrasound on Renal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alper Mengi (Other Government)
Responsible Party: Sponsor-Investigator, Alper Mengi, M.D., Physiatrist, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-99-21/10
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Ultrasound Therapy; Complications; Low Back Pain
Keywords: Chronic Pain; physiotherapy; renal function
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic ultrasound group (Active Comparator): The patients will be treated with superficial heating, transcutaneous electrical nerve stimulation, exercise therapy and therapeutic ultrasound over the paravertebral low back region.
  Interventions: Other: physiotherapy modalities
- therapeutic ultrasound untreated group (Other): The patients will be treated with superficial heating, transcutaneous electrical nerve stimulation, exercise therapy over the paravertebral low back region.Therapeutic ultrasound will not be applied to this group.
  Interventions: Other: physiotherapy modalities

INTERVENTIONS:
Other: physiotherapy modalities — The physiotherapy modalities will be applied for five sessions a week for 3 weeks.
  The all patients will be treated with superficial heating (the moist heat pack will be applied to the patient's lower back for 20 minutes) , transcutaneous electrical nerve stimulation(frequency of 100 Hz, pulse duration of 100 μs, sensory-level amplitude was applied for 25 minutes) , exercise therapy (consisting of flexion, extension, stretching, mobilisation, and postural exercises performed for approximately 25 minutes ) .
  In addition to these therapies, continuous therapeutic ultrasound treatment will be applied to patients in first group for 10 minutes; frequency of 1 megahertz, intensity of 1.5 W/cm2, effective irradiation area of the transducer head 5 cm2 .

SUMMARY:
This study evaluates whether therapeutic ultrasound (TUS) treatment applied to lumbar region with chronic low back pain affect renal function.

DETAILED DESCRIPTION:
Low back pain is a common problem and there are many treatments for chronic low back pain, including TUS. Investigators routinely observed increased blood creatinine and urea levels in some of patients who received TUS.

Half of patients will receive TUS treatment for low back pain while the other half will not receive. The patients will be evaluated at baseline and the end of the treatment . The serum creatinine, serum cystatin C, 24-hour urine creatinine, creatinine clearance, 24-hour urine microalbumin and microprotein, urine volume, and GFR will be measured at each evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 65 years
* with chronic mechanical low back pain for at least 3 months
* with glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m2, as calculated using the Modification of Diet in Renal Disease formula .

Exclusion Criteria:

* history of lumbar surgery
* having inflammatory low back pain
* having pregnancy
* having active infection
* history of malignancy
* having coagulation disorder
* having a cardiac pacemaker
* having heart failure
* having uncontrolled hypertension or hypotension
* having active psychiatric disease
* presence of skin diseases on low back pain
* taking medicines for low back pain during the physical therapy treatment (except for paracetamol)
* taking a new drug for another disease or undergoing a dose change for a drug taken during the course of physiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Concentration of serum creatinine | 1 day
  To measure the serum creatinine levels, 5 mL of venous blood will be collected in a tube containing a gel separator and clot activator in the morning after a 12-hour fast. Serum creatinine will be measured in an autoanalyser.
Value of 24-hour urine creatinine | 1 day
  After the first urine sample of the first day was discarded, 24-hour urine samples will be collected, including the first of the next day. The 24-hour urine samples will be analysed on the day of collection, and will be analysed using colorimetric method in an autoanalyser.
Value of creatinine clearance | 1 day
  Creatinine clearance will be calculated with the following formula:
  Urine creatinine (mg/dL) × urine volume (mL)/serum creatinine (mg/dL) × 1440.
glomerular filtration rate | 1 day
  Glomerular filtration rate will be as calculated using the Modification of Diet in Renal Disease formula. (GFR (mL/min/1.73 m²) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
Concentration of serum cystatin C | 1 day
  To measure the cystatin-C levels, 5 mL of venous blood will be collected in a tube containing a gel separator and clot activator in the morning after a 12-hour fast. Serum cystatin C will be determined using a sandwich enzyme immunoassay kit.
Value of 24-hour urine microalbumin | 1 day
  After the first urine sample of the first day was discarded, 24-hour urine samples will be collected, including the first of the next day. The 24-hour urine samples will be analysed on the day of collection, and will be analysed using immunoturbidimetric method in an autoanalyser.
Value of 24-hour urine microprotein | 1 day
  After the first urine sample of the first day was discarded, 24-hour urine samples will be collected, including the first of the next day. The 24-hour urine samples will be analysed on the day of collection, and will be analysed using colorimetric method in an autoanalyser.

IPD SHARING:
Plan to Share IPD: No